CLINICAL TRIAL: NCT04398758
Title: Prospective, Randomized, Non-treatment-controlled, Investigator-blinded, Multicenter Study on the Prophylaxis of Early Childhood Symptoms of Atopic Dermatitis in High-risk Children by Continuous Application of a Moisturizing Barrier-stabilizing Skin Cream
Brief Title: Moisturizer Mediated Prevention of Symptoms of Atopic Dermatitis in Early Childhood
Acronym: MOPAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOPAD; 2018-004762-33 (EudraCT Number)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis; Infant, Newborn
Keywords: Skin care; Prevention; Risk factor; Interventional study; Multicentric
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, non-treatment-controlled, investigator-blinded, multicenter, 2-arm parallel group study (main phase: from inclusion until 6 months of age with treatment group and control group (without treatment) according to 1:1 randomisation; follow-up phase: 6-12 months of age in which only half of the children from the treatment group is treated according to initial 1:1 randomisation)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Children of the treatment group receive the cream "SanaCutan Basiscreme". The cream's main ingredients are white soft paraffin and liquid paraffin and it is already approved for the treatment of several skin diseases due to its skin care effect.
  Interventions: Drug: SanaCutan Basiscreme
- Control group (No Intervention): Children of the control group should avoid regular skincare applications. Skincare is not prohibited, however, it is recommended to use products only in urgent cases.

INTERVENTIONS:
Drug: SanaCutan Basiscreme — In this study, the SanaCutan Basiscreme will be used as a cream for twice daily application on the whole body (eyes and mucous membranes have to be omitted) for a duration of 6 months (main phase) or 12 months (main + follow-up phase) or less (if the child develops atopic dermatitis).
  Arms: Treatment group

SUMMARY:
In this study, it will be investigated if symptoms of atopic dermatitis of children with high familial risk will be delayed beyond the 6th or even 12th month of life by applying the SanaCutan Basiscreme.

DETAILED DESCRIPTION:
Enrolled healthy newborns with high risk for atopic dermatitis will be 1:1 randomised into treatment and control group. The treatment group receives the SanaCutan Basiscreme for twice daily skin application until the age of 6 months (main phase; half of them until the age of 12 months (main + follow-up phase)), whereas the control group should avoid skin care products. Guardians of both groups are requested to document all applied skin care products in a diary. In regular visits at the study sites, a blinded physician investigates the skin of the children. In case of an atopic dermatitis (= atopic dermatitis has to be diagnosed in at least two visits with an interval of at least four weeks), the severity will be examined (SCORAD) and the treatment with SanaCutan Basiscreme will be terminated. All children will be followed up until the age of 6 months (end of main phase). This is the time when a blood test will be conducted to determine sensitization against food and inhalant allergens and total IgE. If children do not develop an atopic dermatitis in the main phase, the study continues until they receive the diagnosis (up to a maximum of 12 months, end of follow-up phase).

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns (male or female)
* Age < 3 weeks (≤ 21st day of life)
* High familial risk of atopic dermatitis in the form of at least one first-degree relative (parent or sibling) with a medically diagnosed atopic dermatitis in the medical history
* Written consent of all guardians

Exclusion Criteria:

* Acute or chronic diseases
* Acute fever (> 38.5 °C)
* Severe congenital malformations
* Hydrops fetalis
* Immunodeficiency (any kind)
* Severe genetic skin diseases or skin conditions that make the use of skin creams unsuitable
* Corticoid or calcineurin inhibitor use or Ciclosporin intake
* Preterm birth (< 37 weeks)
* Known hypersensitivity to one of the ingredients of the SanaCutan Basiscreme
* Restricted legal capacity of the guardians
* Inability of the guardians to understand the study instructions
* Obvious unreliability or lack of cooperation of the guardians
* Known alcohol, medicine or drug dependency of the guardians
* Dependence of the child or guardians on the sponsor or the investigator
* Previous participation in another clinical trial (since birth)
* Previous participation in this study

Max Age: 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of children with atopic dermatitis at 6 months of age | 0-6 months of age
  A confirmed atopic dermatitis is present if an atopic dermatitis is diagnosed in at least 2 examinations at intervals of at least 4 weeks (preliminary diagnosis + proof of chronification).
  The primary objective is achieved when the cumulative incidence of children with atopic dermatitis in the treatment group at 6 months of age is significantly lower than in the control group without predetermined treatment (p < 0.05).

SECONDARY OUTCOMES:
Cumulative incidence of children with atopic dermatitis at the age of 12 and 16 weeks and 9, 12 and 6-12 months | 0-12 months of age
Cumulative incidence of children with preliminary diagnosis of atopic dermatitis (regardless of whether chronification is confirmed) at 12 and 16 weeks and 6, 9 and 12 months | 0-12 months of age
Time to onset of atopic dermatitis at the age of 0-6, 6-12 and 0-12 months | 0-12 months of age
Cumulative incidence and frequency of children with xerosis at the age of 6 and 12 months | 0-12 months of age
Cumulative incidence and frequency of children with signs of itching at 6 and 12 months of age | 0-12 months of age
Cumulative incidence and frequency of children with other types of eczema at 6 and 12 months of age | 0-12 months of age
Severity of atopic dermatitis at the time of detection of (confirmed) atopic dermatitis up to the age of 12 and 16 weeks and 6, 9 and 12 months | 0-12 months of age
  Method: SCORAD (SCORing Atopic Dermatitis; 0-104 points; higher score indicates a more severe atopic dermatitis)
Frequency of sensitization to food allergens (according to Fx5 test + hazelnut) and to inhalation allergens (according to Sx1 test) and total IgE at the age of 6, 9 and 12 months | 0-12 months of age
  Positive/negative of Fx5 test and Sx1 test and - in case of a positive result - on a single allergen basis (with specific IgE value). The measures of sensitization and total IgE are performed for all children at the age of 6 months and again for children in the follow-up phase, if they are diagnosed with atopic dermatitis in this period of time.
Adverse events: overall frequency, type, severity, causality, with frequencies, separate presentation of local reactions up to the age of 6 and 12 months | 0-12 months of age
Drop-outs (with reasons) up to the age of 6 and 12 months | 0-12 months of age
Compliance regarding the use of the investigational medicinal product in the treatment group up to the age of 6, 12 and 6-12 months | 0-12 months of age
Compliance regarding the use of other skin care products (not investigational medicinal product) in both groups up to the age of 6, 12 and 6-12 months | 0-12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Beyer, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (10):
- Germany (10):
  - Gemeinschaftspraxis Bauer, Gilb, von Bentzel, Augsburg
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Universitätsmedizin, Berlin
  - Evangelisches Klinikum Bethel, Bielefeld
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - St. Marien-Hospital, Bonn
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Barmherzige Brüder Klinik St. Hedwig, Regensburg
  - Gemeinschaftspraxis für Kinder- und Jugendmedizin, Tuttlingen
  - Marien Hospital Wesel, Wesel

IPD SHARING:
Plan to Share IPD: No